CLINICAL TRIAL: NCT05306730
Title: Echocardiography by Non-cardiologist in Early Management of Patients With Chest Pain
Acronym: ENDEMIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Defence, Faculty of Military Health Sciences (Other)
Responsible Party: Principal Investigator, Petr GRENAR, MD, Principal Investigator, University of Defence, Faculty of Military Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-0001-9433-296X
Record Dates: First submitted 2022-02-14; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Cardiology; Acute Coronary Syndrome; Echocardiography
Keywords: Echocardiography; Point-of-care ultrasound
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOCUS group (Experimental): Group of patients with chest pain undergoing FOCUS ( Focused Cardiac Ultrasound ).
  Patients with odd registration number.
  Interventions: Device: ECHOcardiography, Point-of-Care UZ
- Non-FOCUS group (Active Comparator): Patients with even registration number.
  Interventions: Device: ECHOcardiography, Point-of-Care UZ

INTERVENTIONS:
Device: ECHOcardiography, Point-of-Care UZ — Emergent echocardiography is reproducible method providing clinically significant information during primary survey of acute cardiovascular diseases. Possible benefit is the risk stratification of acute non-stemi coronary syndromes and differentiation from other serious conditions, such as pulmonary embolism or aortic dissection. The aim of interest is to consider riscs and benefits of the ultrasound of heart done by non-cardiologist after standardized course.

SUMMARY:
The aim of the study is to find out the benefit of echocardiography, which is performed by a physican without a cardiological or radiological specialty. In this case the echocardiography is used in the first contact with a patient with chest pain of unclear etiology. Possible benefit is rapid risk stratification of acute non-stemi coronary syndromes and differentiation from other serious conditions, such as pulmonary embolism or aortic dissection.

DETAILED DESCRIPTION:
Emergent echocardiography is reproducible method providing clinically significant information during primary survey of acute cardiovascular diseases. Possible benefit is the risk stratification of acute non-stemi coronary syndromes and differentiation from other serious conditions, such as pulmonary embolism or aortic dissection.

Step one - Education in Cardiac ultrasound. All physicians involved in ENDEMIC study have to undergo education program of heart ultrasonography. This curriculum fulfills BSE level one requirements. Candidates of this program have to make a defined number of ECHOcardiography studies under supervisor control. Every curriculum is finished by exam.

Step two - FOCUS in clinical practise Patients with chest pain are randomized into two groups by the even-odd rule.

Inclusion Criteria:

Chest pain ( Cardiovascular ethiology possible depends on anamnesis, physical examination and ECG ) Higher age than 18

Exclusion Criteria:

STEMI Pacemaker / ICD Pregnancy Performance status 4 ( Zubrod scale ) Informed Consent unsigned Prisoners

Step Three - Evaluation

Aims.:

Compare time to make a decision in these groups Compare time of stay at emergency department in these groups Compare time to invasive coronary angiography and revascularization (if available) Compare time to hospital dimission Occurrence of MACE in following 30 days

ELIGIBILITY:
Inclusion Criteria:

* Chest pain ( Cardiovascular ethiology possible depends on anamnesis, physical examination and ECG )
* Higher age than 18

Exclusion Criteria:

* STEMI
* Pacemaker / ICD
* Pregnancy
* Performance status 4 ( Zubrod scale )
* Informed Consent unsigned
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Time of patient stay at Emergency Department | 24 hours
  Time from initial contact with patient to patient discharge or hospital admission (minutes)

SECONDARY OUTCOMES:
Time of stay at hospital | 28 days
  Time from hospital admission to hospital discharge (hours)
Major adverse cardiovascular events | 30 days
  Major adverse cardiovascular events are defined as composite endpoint of cardiovascular death, nonfatal myocardial infarction or unscheduled hospitalization due to cardiovascular disease (percent of patients in study groups).

OTHER OUTCOMES:
Time to Coronary Angiography | 365 days
  Time from initial contact to coronary angiography (days)
Accuracy of thoracic ultrasound exam provided by non-cardiologist | 30 days
  All echocardiography records will be revised by skilled echocardiographist to assess the accuracy of performed examinations. All missed or erroneous finding resulting in alteration of patient management (especially wall motion abnormity, valvular disease and pericardial effusion) will be calculated. (quantity of erroneous or missed findings per record)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Jakl, assoc.prof., Study Director — University of Defense, Faculty of Military Health Sciences, Czech Republic; Petr Grenar, MD, Principal Investigator — University of Defense, Faculty of Military Health Sciences, Czech Republic

IPD SHARING:
Plan to Share IPD: Yes
To be shared:
  * baseline characteristics of study population
  * data related to primary and secondary endpoints
Supporting Information: Study Protocol, CSR
Time Frame: Available 1 year after completing the study, for at least 10 years
Access Criteria: Contact principal investigator

REFERENCES:
- [Derived] Grenar P, Jakl M, Medilek K, Novy J, Koci J, Vanek J, Cermakova M, Horacek JM, Pudil R. Effect of point-of-care echocardiography by noncardiologists on patient management in acute chest pain. Intern Emerg Med. 2025 Nov 24. doi: 10.1007/s11739-025-04198-6. Online ahead of print. PMID 41284127
- [Derived] Grenar P, Novy J, Medilek K, Jakl M. Point-of-Care Cardiac Ultrasound Training Programme: Experience from the University Hospital Hradec Kralove. Emerg Med Int. 2024 Jan 6;2024:9974284. doi: 10.1155/2024/9974284. eCollection 2024. PMID 38222095